CLINICAL TRIAL: NCT07131332
Title: Mindfulness Based Eating and Awareness Training for Post-bariatric Surgery Patients: A Mixed Methods Outcome Study
Brief Title: Mindfulness-Based Eating Awareness Training for Post-bariatric Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Susan Wnuk, Principal Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-5105; 19-5105 (Other: University Health Network)
Record Dates: First submitted 2025-08-04; First posted 2025-08-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Eating Behaviors
Keywords: mindfulness; overeating; metabolic and bariatric surgery; mindful eating; adults
MeSH Terms: conditions — Feeding Behavior; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindful eating group (Experimental): Behavioral group intervention involving 8, 2-hour long sessions
  Interventions: Behavioral: Mindful eating group

INTERVENTIONS:
Behavioral: Mindful eating group — Behavioral group intervention involving 8, 2-hour long sessions

SUMMARY:
The goal of this clinical trial was to see if learning and practicing mindful eating in a group was helpful for people who had bariatric surgery. The main questions it aims to answer are:

1. Does learning and practicing mindful eating help decrease overeating, improve mood, decrease anxiety, and lead to other similar changes?
2. What do people who participated in a mindful eating group find helpful and hindering about it?

Participants were asked to:

* take part in an 8-week mindful eating group
* complete questionnaires before the group started and after it ended, about their eating habits, mood, anxiety and other similar issues
* complete a questionnaire right after each session asking them what they found helpful and hindering about that session

DETAILED DESCRIPTION:
BACKGROUND: Bariatric surgery, specifically the roux-en-y gastric bypass and gastric sleeve, has been conducted at the University Health Network Surgery Program (UHN-BSP) since late 2009. Weight loss through bariatric surgery is associated with the improvement or resolution of medical comorbidities as well as improvements in patient-reported quality of life. Bariatric surgery is also more successful than other weight loss methods in maintaining weight loss. Therefore, weight regain is of primary concern in this population. Psychiatric factors associated with weight regain include binge eating, lack of control over food urges and a greater number of psychiatric disorders.

Mindfulness meditation techniques may address many of the factors related to disordered eating that contributes to weight regain, including distressing emotions and cognitive distortions. Mindfulness training involves purposeful and sustained attention to thoughts, emotions and bodily sensations. This encourages the recognition of and improved ability to tolerate painful emotions without engaging in problematic behavior like overeating. Mindfulness is a well-validated intervention for psychological and medical problems in other patient populations, including anxiety, depression, stress. Mindfulness-Based Eating Awareness Training (MB-EAT) is a group program developed by Kristeller and colleagues that integrates mindfulness meditation and eating meditation with didactics about healthy eating.

Mindfulness and mindful eating practice may help individuals better recognize and respond to feelings of hunger and fullness. Bariatric surgery patients tend to have a history of multiple weight-loss diet attempts. These diets usually emphasize rules for how much, when and what to eat that paradoxically lead to the loss of one's ability to recognize, accept or respond to internal cues of hunger, taste, satiety, and fullness. Studies that that investigated mindful eating interventions for bariatric surgery patients indicate that they improve eating behavior, emotion regulation, and depression. The investigators conducted one of these studies and found that depression and binge eating significantly decreased from pre to post intervention and emotion regulation significantly improved.

OBJECTIVES:

Primary Objective: To quantitatively investigate the effectiveness of MB-EAT in enhancing psychological functioning as an adjunct treatment to the usual standard of care in the 40 bariatric surgery patients who participated in MB-EAT groups.

Secondary Objective: To qualitatively better understand participants' reactions to MB-EAT, specifically perceptions of helpful and unhelpful aspects, via written comments and ratings that were provided at the end of each session.

HYPOTHESES:

Primary Hypothesis (quantitative): The investigators expect that participants will show improvements in psychological functioning from pre to post-MB-EAT.

Secondary Hypothesis (qualitative): Participants will identify helpful and hindering aspects of MB-EAT in their written feedback after each session.

Outcome Measures (quantitative): The primary outcome measures are changes in self-reported eating pathology, depression, anxiety, interoceptive awareness, mindfulness.

Outcome Measure (qualitative): Identification of helpful and hindering aspects of the session just completed.

INCLUSION/EXCLUSION CRITERIA:

Inclusion criteria:

1. Pre and post-bariatric surgery patient enrolled at the UHN-BSP who participated in one of four MB-EAT groups in 2015 and 2016.

Exclusion criteria: None.

INTERVENTION: Eight sessions of MB-EAT delivered once per week over the course of 8 weeks, based on a protocol developed by Kristeller et al. with minor modifications to accommodate the typical dietary restrictions encountered by post-surgery patients. For example, due to abdominal discomfort experienced by post-surgery patients when consuming sugar and fat, sugar-free/fat-free food items were made available for mindful eating exercises that involve sweet foods. Each session was two hours in length. The primary emphasis of MB-EAT is to teach and facilitate mindfulness exercises to help participants gain greater control over their eating. Didactics about healthy eating were provided in addition to instruction in a cognitive behavioral therapy exercise that analyzes problem eating episodes. Homework included daily meditations, mindful eating exercises and occasional worksheets.

MB-EAT groups were co-facilitated by two of three clinicians who work in the TWH-BSP: Susan Wnuk, Ph.D., C. Psych., a clinical psychologist; Chau Du, M.Sc., a psychometrist, and Katie Warwick, R.D. a dietitian All facilitators completed MB-EAT facilitator training and provided clinical care in the UHN-BSP for between 5-7 years.

METHOD

1. Quantitative measures: Participants completed the self-report measures provided by the investigators immediately prior to the start of the first session (baseline) and at the end of the 8th session (week 8).
2. Qualitative measures: Participants completed the self-report qualitative measure provided by the investigators immediately after the completion of all 8 sessions. Thus, data were collected weekly starting at baseline through to week 8.

ELIGIBILITY:
Inclusion Criteria

* Any patient enrolled in the University Health Network Bariatric Surgery Program
* Able to speak, read and write English

Exclusion Criteria:

- Inability to speak, read and write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Binge Eating Scale | Immediately prior to the start of the first MB-EAT session (baseline) and at the end of the 8th session (8 weeks later)
  Self-report questionnaire of eating behaviour typical of binge eating. It contains 16 items and responses for each item range from 1-4. The minimum score is 0 and the maximum score is 46. Higher scores indicate more binge eating.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 | Immediately prior to the start of the first MB-EAT session (baseline) and at the end of the 8th session (8 weeks later).
  Self-report questionnaire of depressive symptoms. It contains 9 items and responses for each item range from 0-3. The minimum total scale score is 0 and the maximum score is 27. Higher scores indicate more depressive symptoms.
Generalized Anxiety Disorder 7 | Immediately prior to the start of the first MB-EAT session (baseline) and at the end of the 8th session (8 weeks later).
  Self-report questionnaire of anxiety symptoms. It contains 7 items and responses for each item range from 0-3. Total scale scores range from 0-21. Higher scores indicate more anxiety symptoms.
Five facets of mindfulness questionnaire | Immediately prior to the start of the first MB-EAT session (baseline) and at the end of the 8th session (8 weeks later).
  Self-report questionnaire of traits associated with mindfulness. It contains 39 items and responses on each item range from 1-5. Total scores range from 39-195. Higher scores indicate more mindfulness.
Multidimensional Assessment of Interoceptive Awareness | Immediately prior to the start of the first MB-EAT session (baseline) and at the end of the 8th session (8 weeks later).
  Self-report questionnaire of interoceptive awareness. It contains 32 items and response range from 0-5. The total scale score ranges from 0-185. Higher scores indicate greater interoceptive abilities.
Helpful Aspects of Therapy Form | Immediately after the completion of each of 8 MB-EAT sessions from baseline (week 1) and weekly until week 8.
  Self-report questionnaire identifying helpful and hindering aspects of the session just completed. It contains 7 main items (1-5) and 4 sub-items (6a, 6b, 7a, 7b) that elicit subjective written responses and numerical ratings. Items 1, 2, 4, 5, 6b and 7b elicit subjective responses about why aspects of the session were helpful or hindering. Item 3 rates the helpfulness of the first identified helpful event on a scale of 0-9: 1=extremely hindering to 9=extremely helpful. Scores range from 1-9. Item 6 asks whether a second helpful event occurred. If yes, 6a rates the helpfulness of the second identified event from 1-4: 1= slightly helpful to 9=extremely helpful. Scores on this item range from 1-4. Item 6b describes what made this event helpful. Item 7 asks whether a hindering event occurred. If yes, item 7a rates the extent from 1=extremely hindering to 4=slightly hindering. Scores range from 1-4. There is no total score computed for this measure.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Wnuk, S.M., Du, C.T., Van Exan, J. et al. Mindfulness-Based Eating and Awareness Training for Post-Bariatric Surgery Patients: a Feasibility Pilot Study. Mindfulness 9, 949-960 (2018).
- [Background] Chacko SA, Yeh GY, Davis RB, Wee CC. A mindfulness-based intervention to control weight after bariatric surgery: Preliminary results from a randomized controlled pilot trial. Complement Ther Med. 2016 Oct;28:13-21. doi: 10.1016/j.ctim.2016.07.001. Epub 2016 Jul 12. PMID 27670865
- [Background] Kristeller JL, Wolever RQ. Mindfulness-based eating awareness training for treating binge eating disorder: the conceptual foundation. Eat Disord. 2011 Jan-Feb;19(1):49-61. doi: 10.1080/10640266.2011.533605. PMID 21181579
- [Background] Goldberg SB, Tucker RP, Greene PA, Davidson RJ, Wampold BE, Kearney DJ, Simpson TL. Mindfulness-based interventions for psychiatric disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2018 Feb;59:52-60. doi: 10.1016/j.cpr.2017.10.011. Epub 2017 Nov 8. PMID 29126747
- [Background] Chesler BE. Emotional eating: a virtually untreated risk factor for outcome following bariatric surgery. ScientificWorldJournal. 2012;2012:365961. doi: 10.1100/2012/365961. Epub 2012 Apr 1. PMID 22566765
- [Background] Rutledge T, Groesz LM, Savu M. Psychiatric factors and weight loss patterns following gastric bypass surgery in a veteran population. Obes Surg. 2011 Jan;21(1):29-35. doi: 10.1007/s11695-009-9923-6. Epub 2009 Jul 15. PMID 19847571
- [Background] White MA, Kalarchian MA, Masheb RM, Marcus MD, Grilo CM. Loss of control over eating predicts outcomes in bariatric surgery patients: a prospective, 24-month follow-up study. J Clin Psychiatry. 2010 Feb;71(2):175-84. doi: 10.4088/JCP.08m04328blu. Epub 2009 Oct 20. PMID 19852902
- [Background] Mitchell JE, Lancaster KL, Burgard MA, Howell LM, Krahn DD, Crosby RD, Wonderlich SA, Gosnell BA. Long-term follow-up of patients' status after gastric bypass. Obes Surg. 2001 Aug;11(4):464-8. doi: 10.1381/096089201321209341. PMID 11501356